CLINICAL TRIAL: NCT04282876
Title: Influence of Hormone Treatment in Radiation Therapy for Bladder Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Jørgen Bjerggaard Jensen, Professor, Aarhus University Hospital
Other Study IDs: 1-10-72-272-19
Record Dates: First submitted 2020-02-19; First posted 2020-02-25 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Bladder Cancer; Radiation Therapy Complication; Quality of Life
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bladder biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Degarelix: Patients undergoing radiation therapy for bladder cancer while also being treated with Degarelix (androgen deprivation therapy)
  Interventions: Drug: Degarelix
- Control: Patients undergoing radiation therapy for bladder cancer with or without simultanous treatment with androgen deprivation therapy (not Degarelix)

INTERVENTIONS:
Drug: Degarelix — Patients receiving Degarelix
  Groups: Degarelix

SUMMARY:
Bladder cancer is often treated with cystectomy or radiation therapy. Following radiation therapy patients will often have severe side effects from the treatment. Studies have suggested that simultanously treatment with androgen deprivation therapy during radiation therapy may be able to proctect stemcells in the bladder, thus improving tissue recovering post-radiation, which would result in improved bladder compliance following the treatment and ultimately result in fewer side effects and overall improved patient quality of life.

DETAILED DESCRIPTION:
Bladder cancer (BC) is one of the most frequent cancers in the world and more common in men than female. Gender-related factors may be involved in the pathogenesis of BC.

Studies have suggested that androgen-receptors may be present in the bladder and potentially involved in BC aetiology, thus making BC susceptible for androgen deprivation therapy (ADT).

Currently treatment for BC includes surgery or radiation therapy. ADT include Degarelix, which besides decreasing testosterone, has been shown to reduce the occurrence of BC in rats and promote stem cell recovery following radiation therapy.

Hypothesis ADT will lower the incidence of BC, and the prognosis of BC will vary depending on the type of ADT used. Furthermore Degarelix administered during radiation therapy for BC will reduce the degree of fibrosis in the bladder thus decreasing adverse side effects.

Methods A cohort of patients treated with ADT for PC will be compared to two cohorts of age-matched men with and without PC both without ADT. The incidence of BC will be recorded for every group. Furthermore the cohort of patients with PC and ADT will be divided into subgroups, depending of the type of ADT they have received and the degree of deprivation. They will be compared in terms of incidence and prognosis of BC.

Finally, a small pilot study will be conducted to investigate the effect of Degarelix when administered during radiation therapy for BC.

Perspectives This will be one of the largest studies to investigate the potential influence of sex hormones in the development and prognosis of BC and potentially lead to new treatment options and possibly a new way of reducing radiation side effects.

ELIGIBILITY:
Inclusion Criteria:

* T2-T4 bladder cancer
* radiation therapy
* able to fill out questionnaires
* signed informed consent

Exclusion Criteria:

* KAD prior to TUR-B
* dementia or other cognitive impairment
* metastatic disease

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: Males with invasive bladder cancer, treated with radiation therapy.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-02-19 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Bladder fibrosis | 3 months after radiation
  Fibrosis of the bladder determined by bladder biopsy estimated by number of fibrotic fibers on IHC staining

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No